CLINICAL TRIAL: NCT04222829
Title: Observational Study on Effectiveness of Megadose Shinbaro Pharmacopuncture for Patients With Chronic Shoulder Pain Due to the Shoulder Diseases
Brief Title: The Effectiveness of Megadose Shinbaro Pharmacopuncture for Patients With Chronic Shoulder Pain
Status: Terminated | Type: Observational
Why Stopped: low participate rate
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2019-09
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Shoulder Joint Disorder
Keywords: Shoulder joints; Shinbaro pharmacopuncture; Megadose shinbaro pharmacopuncture; Chronic shoulder pain; Shoulder pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Megadose Shinbaro Pharmacopuncture Group: The Megadose Shinbaro Pharmacopuncture group who are treated with korean medical treatment including Megadose Shinbaro Pharmacopuncture will be evaluated on first, second, third visit and 2weeks after baseline. And the patients will receive telephone inquires after 3months from the baseline.
  The Korean medical treatment includes acupuncture, chuna and Korean herbal medicine.
  Interventions: Procedure: Megadose Shinbaro Pharmacopuncture
- Control Group: The control group who are treated with Korean medical treatment not including Megadose Shinbaro Pharmacopuncture will be evaluated on first, second, third visit and 2weeks after baseline. And the patients will receive telephone inquires after 3months from the baseline.
  The Korean medical treatment includes acupuncture, chuna and Korean herbal medicine.

INTERVENTIONS:
Procedure: Megadose Shinbaro Pharmacopuncture — Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints.
  Shinbaro is a refined herbal formulation used to treat inflamed lesions and bone diseases.
  Groups: Megadose Shinbaro Pharmacopuncture Group

SUMMARY:
This study is a prospective, case-control observational trial. The investigators will compare the Megadose Shinbaro Pharmacopuncture group to the control group to analyze the effectiveness of shoulder Megadose Shinbaro Pharmacopuncture.

DETAILED DESCRIPTION:
Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints.

Shinbaro is a refined herbal formulation used to treat inflamed lesions and bone diseases.

This treatment is known to be an important part of Korean medicine treatment. However, there has been no specific value for the effect of this treatment.

Therefore, The investigators conducted observational trial to analyze the effectiveness of Megadose Shinbaro Pharmacopuncture on shoulder. From Dec 2019, The investigators will collect 80 patients with Chronic shoulder pain on both or each shoulder with the numeric rating scale(NRS) over 4.

The investigators will compare pain, dysfunction, quality of life and satisfaction of patients who are treated with Korean medical treatment including Megadose Shinbaro Pharmacopuncture and patients who are treated with Korean medical treatment not including Megadose Shinbaro Pharmacopuncture.

For these two groups, The investigators will compare NRS(Numeric Rating Scale), Visual Analogue Scale(VAS), Range Of Motion(ROM), Shoulder Pain and Disability Index(SPADI), Patient Global Impression of Change (PGIC) and EuroQol 5-Dimension (EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

* Patients with NRS ≥ 4 for shoulder pain over 3weeks
* Patients aged 19-70 years on the date they sign the consent form.
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients who have been diagnosed with a severe disease that may cause shoulder pain,
* Patients with progressive neurological deficit or with serious neurological symptoms caused by spinal cord compression.
* Patients who visited a hospital in pain caused by a traffic accident.
* Patients with a severe mental illness.
* Patients who are difficult to complete the research participation agreement

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated in Haeundae Jaseng Korean Medicine Hospital
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale of shoulder pain | At 2 weeks
  The extent of shoulder pain and discomfort was assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their shoulder pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Visual Analogue Scale of shoulder pain | At screening, baseline, 2 weeks and through study completion, an average of 3 month
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end. Higher scores mean a worse outcome
Shoulder mobility on the Shoulder ROM | At baseline, 2 weeks and through study completion, an average of 3 month
  Shoulder ROM was measured in six directions (Flexion, Extension, Abduction, Adduction, Right rotation, Left rotation) with goniometer.
Shoulder Pain and Disability Index questionnaire of shoulder pain and disability | At baseline, 2 weeks, 3 months
  SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. Higher scores mean a worse outcome
Patient Global Impression of Change | At baseline, 2 weeks, 3 months
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
EuroQol 5-Dimension | At baseline, 2 weeks, 3 months
  The EQ-5D-5L is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, The investigators will use the Korean version of the EQ-5D-5L, which has been demonstrated to be valid.
Number of Participants with Adverse events | Through study completion, an average of 3 month
  Adverse events(AE) Physicians will monitor and record any unexpected or unintended patient reaction to integrative korean medicine at each visit. Adverse events (AEs) associated with integrative korean medicine will include, but not be limited to, AEs anticipated from previous reports of korean medicine, and will stay open to all possibilities taking into consideration other potential, unknown AEs.
Numeric Rating Scale of shoulder pain | At screening, baseline, 3 months and through study completion, an average of 3 month
  The extent of shoulder pain and discomfort was assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their shoulder pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Study Chair — Jaseng Medical Foundation
Locations (1):
- Haeundae Jaseng Hospital of Korean Medicine, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided